CLINICAL TRIAL: NCT02009306
Title: Can Nasal Fentanyl and Buccal Midazolam Give Better Symptom Control for Dying Patients When Compared With Standard Subcutaneous Medication? Pilot Randomised Controlled Trial and Qualitative Interview Study.
Brief Title: Nasal Fentanyl and Buccal Midazolam for Dying Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Paul Perkins, Consultant in Palliative Medicine, Gloucestershire Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PecEp1
Record Dates: First submitted 2013-11-18; First posted 2013-12-11 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Terminal Cancer
Keywords: Palliative; Symptom control; Hospice; Opioid; Benzodiazepine
MeSH Terms: interventions — Fentanyl; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PecFent and Epistatus (Experimental): Medication administered by family / carer for symptoms
  Interventions: Drug: PecFent and Epistatus; Drug: Standard subcutaneous medication
- Standard subcutaneous medication (Active Comparator): Standard subcutaneous medication - diamophine and / or midazolam administered by nursing staff
  Interventions: Drug: Standard subcutaneous medication
- Epistatus Alone (Experimental): From 28/11/17 following approval from sponsor, ethics committee and MHRA a 3rd observational arm was introduced:
  Epistatus administered PRN by family / carer for symptoms
  Interventions: Drug: Standard subcutaneous medication; Drug: Epistatus Alone

INTERVENTIONS:
Drug: PecFent and Epistatus — PecFent will be supplied by Archimedes Pharma as two strengths of nasal spray solution at 1000 or 4000 mcg/mL fentanyl (as citrate). One spray contains 100 mcg or 400 mcg fentanyl (as citrate). Each bottle contains 1.55 ml ensuring delivery of 8 sprays of 100 or 400 mcg fentanyl (as citrate). PecFent is a commercially available product and packaging will be in accordance with the manufacturing authorisations (EU/1/10/644/001, EU/1/10/644/002, EU/1/10/644/005, EU/1/10/644/003, EU/1/10/644/004, EU/1/10/644/006).
  Epistatus will be supplied by Special Products Ltd. as buccal solution, packed in bottles containing solution for up to 4 x 1 ml doses, as per "Specials" licence. A pack also includes 4 x oral syringes used to administer the solution to the buccal cavity on either side of the mouth.
  Other Names: Fentanyl and Midazolam
  Arms: PecFent and Epistatus
Drug: Standard subcutaneous medication — Subcutaneous as needed medication will include:
  * Opioids for pain or dyspnoea
    * Diamorphine
    * Oxycodone
    * Fentanyl
  * Benzodiazepine and / or anti-psychotic for agitation
    * Midazolam
    * Levomepromazine
    * Haloperidol Anti-emetic for nausea
  * Cyclizine
  * Metoclopramide
  * Haloperidol
  * Levomepromazine
  * Anti-secretory drug for respiratory secretions
  * Glycopyrronium
  * Hyoscine butylbromide
  * Hyoscine hydrobromide
  Other Names: Subcutaneous opioids and midazolam
Drug: Epistatus Alone — Epistatus will be supplied by Special Products Ltd. as buccal solution, packed in bottles containing solution for up to 4 x 1 ml doses, as per "Specials" licence. A pack also includes 4 x oral syringes used to administer the solution to the buccal cavity on either side of the mouth.
  Other Names: Midazolam
  Arms: Epistatus Alone

SUMMARY:
When patients are dying they become unable to take oral medication and if they develop symptoms (e.g. pain or agitation) they need to be given a subcutaneous injection of medication. If they are at home this requires that a District Nurse is called and it can take a long time (sometimes hours) for the Nurse to arrive. This can be a very stressful time for the patient and family.

There are 2 drug preparations which could potentially be given by family members in the home:

Nasal fentanyl (PecFent) Buccal midazolam (Epistatus) If these preparations helped symptoms this would give much quicker symptom control for patients and might mean the District Nurse visit was not needed.

In advance of a community based randomised trial of these modes of administration, it is important to assess the feasibility of such an approach in terms of carer acceptability and patient tolerability as well as determine appropriate sample sizes and sampling methods. There are 2 work packages which would help assess feasibility of a community trial:

1. An open label randomised controlled trial comparing the use of PecFent with or without Epistatus versus standard subcutaneous breakthrough medication for the management of breakthrough pain (with or without agitation) in dying hospice patients who either remain in the hospice or go home.
2. A qualitative interview study to capture the thoughts of relatives of these patients about the use of these preparations.

DETAILED DESCRIPTION:
This will be an open-label, randomized, controlled feasibility pilot study to evaluate whether using nasal fentanyl (PecFent: 100, 200, 400 or 800 mcg) alone or in combination with buccal midazolam (Epistatus: 2.5, 5 or 10 mg) has the possibility to give better breakthrough symptom control to dying patients when compared with standard subcutaneous medication (Figure 1 A and B).

Each subject and their carers/family members will receive verbal and written information followed by signing of the Informed Consent Forms (ICFs). The study is divided into two arms. In both arms patients will receive standard regular oral or subcutaneous medication for relieving non-breakthrough symptoms. In the standard care arm, patients will receive standard as needed medication (SANM) administered orally, sublingually or subcutaneously for breakthrough symptoms. The experimental arm will consist of two stages: in Stage 1 of the study, PecFent will be given to patients in order to treat breakthrough pain instead of subcutaneous opioids. PecFent will be titrated in order to establish an effective treatment dose to manage pain. SANM administered orally, sublingually or subcutaneously will be used to treat agitation and other symptoms.

After the effective treatment dose of PecFent has been established patients will enter stage 2. Patients will not move to stage 2 if the treatment dose of PecFent is not deemed effective. Stage 2 will test a range of doses of Epistatus in terms of efficacy in treating agitation alone instead of subcutaneous midazolam (or in combination with the effective treatment dose of PecFent for pain and agitation).

SANM will be used to treat other symptoms. Assessment of effectiveness of any as needed medication will be conducted at 30 minutes from administration. If PecFent, Epistatus or a combination of both is ineffective, administration of SANM will be considered. Further opioid cannot be given within one hour but benzodiazepine can be given within 30 minutes as is standard practice in this setting. Thus, patients in the experimental arm will receive symptom relief regardless the efficacy of test drugs.

ELIGIBILITY:
Inclusion Criteria:

Adult hospice in-patients fitting the following criteria will be approached to see if they are willing to participate in the study:

1. diagnosis of terminal cancer and thought to have an estimated prognosis of between 1 and 2 weeks
2. have capacity to consent to participation
3. patients who, in the last 24 hours, have experienced at least one episode of breakthrough pain FOR ARMS 1 OR 2 (RCT) For Arm 3 must have had 1 episode of agitation necessitating the use of a benzodiazepine in the last 24 hours
4. taking 60mg or more of oral morphine (or its equivalent) per 24 hours FOR ARMS 1 OR 2 (RCT) IF taking less than this dose of opioid could be enrolled in Arm 3 (Epistatus alone - change in protocol implemented 28/11/17
5. have carers or family members who would be: willing to give the study medication to the patient likely to be at the hospice at least 50% of the time so that they are likely to be present to administer medication.

Exclusion Criteria:

1. patients / carers / family members who in the opinion of the clinical team would be too distressed by the idea of participation
2. patients with disease of the nasal/buccal mucosa preventing effective absorption of medication
3. families who are unable to administer breakthrough medication e.g. problems with dexterity
4. history of substance abuse - patient or carer / family.
5. people who who might not adequately understand verbal explanations or written information given in English. The pilot is only recruiting 20 patients and Gloucestershire has a only a very small percentage of people who are not English speaking. It has been decided that it is not cost effective to fund translation for this pilot although this information will have to be taken into account when planning a larger study. We will capture information on the numbers of patients that may have been excluded and the languages that might have been needed.
6. Participated in a medicinal trial within the last four months following the guidance from the Association of the British Pharmaceutical Industry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Time to adequate symptom control ('comfortable') from need for breakthrough medication (in minutes) according to patient (where possible), relatives and staff. | 30 minutes
  Data will be captured by patient and/or carer and/or staff with regard to time from need for breakthrough medication (recognition of symptom) to adequate symptom control ('comfortable').

SECONDARY OUTCOMES:
Time (in minutes) from need for breakthrough medication (recognition of symptom) to administration of drug. | 30 minutes
  Data will be captured by patient and/or carer and/or staff with regard to time from need for breakthrough medication (recognition of symptom) to administration of drug.
Need for additional oral or subcutaneous medication | 30 minutes
  Data will be captured by patient and/or carer and/or staff with regard to need for additional oral or subcutaneous medication
Time (in minutes) to recurrence of symptoms according to patient (where possible), relatives and staff | 4 hours
  Data will be captured by patient and/or carer and/or staff with regard to symptoms recurring.
Patient comfort as measured by the modified Palliative care Outcome Scale Symptom list (POS-S) (patient /carer/ staff versions) | 30 minutes
  The modified Palliative care Outcome Scale Symptom list (POS-S) (patient /carer/ staff versions) at approximately the same time daily (depending on when family / carers are likely to be present).
  For this study the Palliative care Outcome Scale Symptom list (known as POS-S) has been modified by removing the question on 'Any other symptoms' and with the addition of the anxiety question from the Integrated Palliative care Outcome Scale (IPOS).
Visual analogue scales for pain and agitation completed by patient (where possible), relatives and staff at baseline (Time 0), 5, 10, 15, 20, 25 and 30 minutes for 1 breakthrough episode per day | 30 minutes
  Visual analogue scales for pain and agitation completed by patient (where possible), relatives and staff at baseline (Time X), time 0 (dose), 5, 10, 15, 20, 25 and 30 minutes (post-dose calculated from time 0) for 1 breakthrough episode per day
Adverse events | 4 weeks after enrolment
  Adverse event information will be collected by research staff.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Perkins, MB BCh FRCP (UK), Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust and
Locations (1):
- Sue Ryder Leckhampton Court Hospice, Cheltenham, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Happy for researchers to contact us once data has been analysed and published

REFERENCES:
- [Derived] Perkins P, Parkinson A, Akyea RK, Husbands E. Nasal fentanyl alone plus buccal midazolam: an open-label, randomised, controlled feasibility study in the dying. BMJ Support Palliat Care. 2020 Sep;10(3):300-303. doi: 10.1136/bmjspcare-2019-002029. Epub 2020 May 6. PMID 32376759